CLINICAL TRIAL: NCT07321743
Title: A Comparative Study Between Stapled and Handsewn Intestinal Anastmosis in Emergency Laparotomy
Brief Title: Emergency Intestinal Anastmosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Reham Zakaria Mohamed Ahmed, lecturer of general surgery, Zagazig University, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 942\31-Dec-2024
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Intestinal Anastomosis
Keywords: stapler; handsewn; anastomotic leakage; intestinal obstruction
MeSH Terms: conditions — Anastomotic Leak; Intestinal Obstruction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stapled group (Active Comparator)
  Interventions: Procedure: emergency intestinal anastmosis surgery
- handsewn group (Active Comparator)
  Interventions: Procedure: emergency intestinal anastmosis surgery

INTERVENTIONS:
Procedure: emergency intestinal anastmosis surgery — cases with intestinal trauma, perforation or intestinal obstruction had emergency laparotomy and intestinal anastmosis was done

SUMMARY:
The goal of this clinical trial is to compare the outcomes of emergency intestinal anastomosis after stapled and handsewn anastmosis. The main question it aims to answer are:

Is stapled intestinal anastmosis is better than handsewn anastmosis in emergency laparotomy?

Participants at surgical emergency unit:

* Had intestinal anastmosis either by stapler or handsewn.
* kept in hospital for follow up and detection of complications like wound infection and leakage.
* Either discharged or managed according to the complications
* Outcomes were compared between the two groups

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to emergency surgery and needed intestinal anastmosis

Exclusion Criteria:

* patients below 18 years old
* immune-compromised patients e.g. corticosteroids therapy, autoimmue disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-12-20 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
intestinal leakage | from one day to two weeks after surgery
  intestinal leakage output calculated in ml by weighing dressing or calculating the drain output

SECONDARY OUTCOMES:
operation time | from incision time to closure (0 to 5 hours)
  operation time in minutes was calculated
bleeding | from one hour to two days after surgery
  bleeding amount was calculated in ml
hospital stay | from one day to one month after surgery
  hospital stay was recorded in days
post-operative pain | from one to three days after after surgery
  pain was evaluated by the visual analogue scale from 1 to 10. score 1 means least painful, score 10 means very painful

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine, Zagazig University, Zagazig, Sharqia Province, Egypt